CLINICAL TRIAL: NCT01876290
Title: Should we Associate Dexamethasone and Ondansetron to Closed-loop Anesthesia to Reduce the Incidence of Postoperative Nausea and Vomiting After Bariatric Surgery?
Brief Title: Dexamethasone and Ondansetron Versus Placebo for Postoperative Nausea and Vomiting
Acronym: Loop-NVPO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2012/14; 2012-001486-32 (EudraCT Number)
Record Dates: First submitted 2013-05-29; First posted 2013-06-12 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Anesthesiology; Complications; Closed-loop
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone and Ondansetron (Experimental): Each patient will receive Dexamethasone and Ondansetron
  Interventions: Drug: Dexamethasone and Ondansetron
- Placebo (Placebo Comparator): Each patient will receive placebo instead of Dexamethasone and Ondansetron
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone and Ondansetron — Comparison between Dexamethasone and Ondansetron and placebo in the prevention of postoperative Nausea and Vomiting
  Arms: Dexamethasone and Ondansetron
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The investigators want to test if it is indicated to associate dexamethasone and ondansetron in obese patients having bariatric surgery under total intra-venous closed-loop anesthesia.

DETAILED DESCRIPTION:
Obese patients having bariatric surgery have frequently postoperative nausea and vomiting (PONV). We want to test if it is indicated to associate dexamethasone and ondansetron in obese patients having bariatric surgery under total intra-venous closed-loop anesthesia.

Two groups to be studied: one will receive 4 mg dexamethasone at the end of the anesthetic induction and 4 mg ondansetron at the end of the surgical procedure, one will receive normal saline.

One hundred twenty consecutive patients meeting the inclusion and exclusion criteria and who give written informed consent to participate in the study will be randomly assigned to one of two experimental groups using a 1:1 ratio.

Patients will be continuously monitored in the post anesthesia care unit (PACU) and the medical floor for a total of 24 hours post operatively. Episodes of nausea, vomiting and administration of rescue therapy for either nausea or vomiting will be recorded and time stamped. In addition, severity of nausea will be evaluated by the patient using a standard verbal response scale (VRS) ranging from 0-10, 0 being no nausea and 10 being severe nausea. Rescue therapy for PONV episodes will consist of 4 mg ondansetron followed by 0.625 mg droperidol if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-75 years
* Scheduled for bariatric surgery under total intra-venous closed-loop anesthesia
* Apfel score equal or greater than 2
* Consenting to participate in the study

Exclusion Criteria:

* Pregnant, breast feeding women
* Allergy
* Contraindication to dexamethasone
* Contraindication to ondansetron
* Contraindication to propofol, remifentanil, morphine, ketoprofen
* Limit to the use of bispectral index

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea or vomiting | 24 hours
  Severe nausea (> to 4 on a 0-10 visual analogue scale) or vomiting

SECONDARY OUTCOMES:
incidence of nausea | one day after anesthesia
  incidence of nausea with delay of occurrence and severity (0-10 visual analogue scale)
incidence of vomiting | one day after anesthesia
  incidence of vomiting with delay of occurrence
rescue treatment | one day after anesthesia
  use of rescue treatment for PONV
pain | one day after anesthesia
  postoperative pain score (0-10 visual analogue scale)
sedation | one day after surgery
  postoperative sedation (0-10 visual analogue scale)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (1):
- Clinique de la Baie des Citrons, Nouméa, France

REFERENCES:
- [Background] Liu N, Chazot T, Hamada S, Landais A, Boichut N, Dussaussoy C, Trillat B, Beydon L, Samain E, Sessler DI, Fischler M. Closed-loop coadministration of propofol and remifentanil guided by bispectral index: a randomized multicenter study. Anesth Analg. 2011 Mar;112(3):546-57. doi: 10.1213/ANE.0b013e318205680b. Epub 2011 Jan 13. PMID 21233500
- [Background] Song JW, Park EY, Lee JG, Park YS, Kang BC, Shim YH. The effect of combining dexamethasone with ondansetron for nausea and vomiting associated with fentanyl-based intravenous patient-controlled analgesia. Anaesthesia. 2011 Apr;66(4):263-7. doi: 10.1111/j.1365-2044.2011.06648.x. PMID 21401538
- [Derived] Bataille A, Letourneulx JF, Charmeau A, Lemedioni P, Leger P, Chazot T, Le Guen M, Diemunsch P, Fischler M, Liu N. Impact of a prophylactic combination of dexamethasone-ondansetron on postoperative nausea and vomiting in obese adult patients undergoing laparoscopic sleeve gastrectomy during closed-loop propofol-remifentanil anaesthesia: A randomised double-blind placebo-controlled study. Eur J Anaesthesiol. 2016 Dec;33(12):898-905. doi: 10.1097/EJA.0000000000000427. PMID 26866433